CLINICAL TRIAL: NCT06363383
Title: A Double-blind Placebo-controlled Phase 1 Study to Evaluate the Safety and Efficacy of MB-001 in Single and Multiple Ascending Doses in Healthy Human Participants
Brief Title: A Phase 1 Study to Evaluate the Safety of an Oral Biologic in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mage Biologics (Industry)
Collaborators: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB-001-101
Record Dates: First submitted 2024-03-29; First posted 2024-04-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: two-stage, single-center, double-blinded, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded using matching placebo capsules containing matching pellets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MB-001 capsules (Experimental): Hard shell capsules for oral use as a single administration or multiple daily administrations over five consecutive days
  Interventions: Biological: MB-001
- Placebo capsules (Placebo Comparator): Matching hard shell placebo capsules for oral use as a single administration or multiple daily administrations over five consecutive days
  Interventions: Biological: MB-001

INTERVENTIONS:
Biological: MB-001 — Oral, delayed release formulation of a biologic drug

SUMMARY:
The goal of this clinical trial is to learn if the oral biologic MB-001 is safe in healthy volunteers. The main questions it aims to answer are:

Is the drug safe when administered orally at increasing doses? Researchers will compare the drug with placebo to see if there are more side effects in those receiving the drug.

Participants will receive a single or five daily doses of the drug or placebo and will be asked to stay in the clinic for five days following the last dose.

DETAILED DESCRIPTION:
This is a two-stage, single-center, double-blinded, randomized, placebo-controlled study evaluating the safety ofMB-001 in healthy adult participants.

The two stages are:

* A single ascending dose (SAD) stage in healthy participants.
* A multiple ascending dose (MAD) stage in healthy participants.

Up to 5 cohorts of healthy adult participants will receive a single oral dose of either MB-001 or placebo. Following a review of all safety data available for the current cohort and any preceding cohorts, the Safety Review Committee (SRC) will decide whether to proceed to the next cohort. The MAD stage in healthy participants will commence once sufficient safety data are available from the SAD stage, after the completion of all SAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to the conduct of any study-related assessment.
2. Adults aged 18 to 65 years, inclusive, at the time of signing the informed consent form (ICF).
3. Body mass index of 18 to 30 kg/m2 , inclusive, at Screening.
4. Estimated glomerular filtration rate > 60 mL/min/1.73m2 at screening, calculated using the Chronic Kidney Disease Epidemiology Collaboration formula.
5. Participants of childbearing potential, fertile male participants, and the female partners of childbearing potential of fertile male participants, must agree to abstain from sexual intercourse or must agree to use highly effective or acceptable methods of contraception from the first dose of study drug until 28 days after the last dose of study drug.
6. Agrees not to donate sperm or ova from first dose of study drug until 90 days or 30 days, respectively, after the last dose of study drug.
7. Willing and able to comply with the study requirements, including remaining at the CRU for the in-house portion of study participation.
8. Agrees not to smoke, vape, or consume tobacco or other nicotine-containing products, from screening until the end of study participation. This includes the use of nicotine patches.
9. Agrees not to consume alcohol from 3 days prior to first dose of study drug until the end of the in-house portion of study participation.
10. Agrees not to consume products containing caffeine or other xanthines from 2 days prior to first dose of study drug until the end of the in-house portion of study participation.
11. Is in good health based on medical history, physical examination, vital signs measurements, safety laboratory tests, and electrocardiograms (ECGs) performed at screening.

Exclusion Criteria:

1. Has any condition that places the participant at significantly increased risk or may compromise the study objectives.
2. Is mentally or legally incapacitated, at screening or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder that would impact study conduct.
3. Has a history of lymphoma, leukemia, or any malignant neoplasms or carcinoma in situ within 5 years prior to screening (except successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix).
4. Regularly consumes more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) within 1 month prior to screening.
5. Has a history of drug or alcohol abuse (defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) within 3 months prior to screening.
6. Females who are pregnant or lactating.
7. For participants of childbearing potential, has a positive pregnancy test at screening or Day -1.
8. Has a QTc > 450 msec for male participants or > 470 msec for female participants at screening or Day -1. NOTE: The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF = QT/(RR^0.33).
9. Has any 12-lead ECG finding at screening or prior to first dose of study drug that may, in the opinion of the Investigator, compromise interpretation of ECGs for cardiac safety assessment or complicate interpretation of events that may occur post dose (e.g., QT not accurately measurable, conduction abnormalities).
10. Has alanine transaminase or aspartate transaminase levels > 1.5 x upper limit of normal (ULN) at screening or Day -1.
11. Has total bilirubin > 1.5 x ULN (isolated bilirubin > 1.5 x ULN is acceptable if total bilirubin is fractionated and direct bilirubin is < 35%) at screening or Day -1.
12. Has a current or chronic history of liver disease. This includes, but is not limited to, hepatitis virus infections, drug- or alcohol-related liver disease, non-alcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the Investigator.
13. Has known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
14. Has a positive test for the presence of HIV, hepatitis C antibody, hepatitis B surface antigen or hepatitis B core antibody at screening or within 3 months prior to first dose of study drug.
15. Has had symptomatic herpes zoster within 3 months prior to first dose of study drug.
16. Has evidence of active or latent tuberculosis (TB) at screening, as documented by QuantiFERON® TB Gold Plus test.
17. Has received treatment with a live, attenuated vaccine within 4 weeks prior to randomization or anticipation of need for such a vaccine during the study period.
18. Has a contraindication to blood sampling or is considered to have insufficient peripheral venous access.
19. Has donated or lost blood or blood products in volumes of 450 mL or more from 30 days prior to first dose of study drug until the end of study participation.
20. Has a history of any known relevant allergy/hypersensitivity or intolerance (including allergy or intolerance to the study medication or its excipients, or to other humanized monoclonal antibodies).
21. Has clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
22. Has a sensitivity to heparin or history of heparin-induced thrombocytopenia.
23. Has a clinically significant infection requiring the use of oral or intravenous anti-infective therapy within 30 days prior to screening.
24. Has abnormal blood pressure, as determined by the Investigator, at screening or Day -1.
25. Has a clinically significant medical condition that, in the investigator's opinion, would preclude participation in the study.
26. Has a positive urine drug screen (including methamphetamine, opiates, cocaine, tetrahydrocannabinol, phencyclidine, benzodiazepines, barbiturates, methadone, tricyclic antidepressants, and amphetamine) at screening or Day -1. Repeat analyses will be allowed if the investigator suspects that there might be false positive results.
27. Has a positive alcohol breath test at screening or Day -1.
28. Has had prior exposure to MB-001.
29. Has participated in a study of any investigational drug, device, biologic, or other agent within 30 days or 5 half-lives prior to signing the ICF, whichever is longer.
30. Has consumed any prescription or over-the-counter medication or herbal/vitamin supplement within 30 days prior to first dose of study drug.
31. Participation in strenuous exercise within 3 days prior to first dose of study drug.
32. Has any history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities, diseases, or genetic conditions. Participants with a remote history of uncomplicated medical events (e.g., uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma) may be enrolled at the discretion of the investigator.
33. Has any clinically significant abnormality identified in the physical examination (including vital signs), laboratory testing, or ECG testing at screening or Day -1. Repeat testing of vital signs to confirm the value is allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | up to day 33 post dosing
  The rate and severity of adverse events occurring from first administration until completion of the study will be collected
Clinically significant changes from baseline in vital signs | up to day 33 post dosing
  Number of participants with clinically significant changes from baseline in vital signs
Clinically significant changes from baseline in physical examination findings | up to day 33 post dosing
  At screening, a complete physical examination will be performed and at subsequent visits, a limited, symptom-directed physical examination will be performed. Any abnormality identified will be recorded either as medical history or as an AE accordingly.
Clinically significant changes from baseline in clinical laboratory assessments | up to day 33 post dosing
  Number of participants with clinically significant changes in laboratory measurements
Clinically significant changes from baseline in ECG parameters | up to day 33 post dosing
  Number of participants with clinically significant changes in ECG parameters

SECONDARY OUTCOMES:
Area under the concentration-time curve | up to 28 days post dosing in the single dose group
  Plasma levels following drug administration will be determined as area under the concentration-time curve
Maximum plasma concentration | up to 28 days post dosing in the single dose group
  The maximum plasma concentration reached after drug administration will be determined
Time to reach observed maximum plasma concentration after administration | up to 28 days post dosing in the single dose group
  The time from drug administration until the maximum plasma concentration is reached will be calculated
Trough concentration | up to day 33 post dosing in the multiple dose group
  The lowest plasma concentrations will be determined after each dosing prior to the next dosing in the multiple dose group

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Spleiss, Study Chair — Mage Biologics
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Placebo data may be shared based on a scientifically acceptable synopsis if in line with ICF